CLINICAL TRIAL: NCT07054996
Title: Investigation of the Effects of Basic Body Awareness Training on Motor Skills, Play Skills, and Social Participation in Children at Risk of Developmental Delay
Brief Title: Investigation of the Effects of Basic Body Awareness Training on Motor Skills İn Children at Risk of Developmental Delay
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, HİLAL DOĞAN, lecturer, Harran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025/083
Record Dates: First submitted 2025-06-26; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Developmental Delay; Body Perception
Keywords: basic body awareness therapy; Motor development; Body perception; Mental rotation; developmental delay
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Basic Body Awareness Group (Experimental): This group will receive basic body awareness training
  Interventions: Other: body awareness therapy
- Play-based Exercise Group (Experimental): An obstacle course will be set up for this group and play-based exercise methods will be implemented.
  Interventions: Other: play-based exercise

INTERVENTIONS:
Other: body awareness therapy — Basic body awareness training will be applied to preschool children in terms of motor development and body perception
  Arms: Basic Body Awareness Group
Other: play-based exercise — Play-based exercise training will be implemented for preschool children by designing games that they enjoy playing, in order to support motor development and body perception.
  Arms: Play-based Exercise Group

SUMMARY:
The aim of this study is to investigate the effects of basic body awareness training on preschool children with developmental delays.

DETAILED DESCRIPTION:
In this study, the effects of basic body awareness training and play-based exercise will be investigated in children with developmental delays. These effects will be evaluated in terms of motor skills, play skills, and social participation

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 6 years attending preschool
* Those who voluntarily agreed to participate in the study

Exclusion Criteria:

* Children with neurological problems
* Children who are uncooperative
* Children receiving speech and language therapy

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
motor development | 1. week- 12. week
  Bruininks-Oseretsky Test of Motor Proficiency. A person can receive a maximum raw score of 72 on the test. A higher score indicates better motor proficiency.
body perception | 1. week- 12. week
  A web-based application will be designed for body perception to help children recognize the parts of their own body using body part images, distinguish between right and left, and measure their reaction speed based on their correct responses to these images

CONTACTS AND LOCATIONS:
Locations (1):
- Milli Eğitim, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD used only for the publication of the results

REFERENCES:
- [Background] Jones RA, Riethmuller A, Hesketh K, Trezise J, Batterham M, Okely AD. Promoting fundamental movement skill development and physical activity in early childhood settings: a cluster randomized controlled trial. Pediatr Exerc Sci. 2011 Nov;23(4):600-15. doi: 10.1123/pes.23.4.600. PMID 22109783